CLINICAL TRIAL: NCT04453787
Title: The Effects of Different Types of Foot Orthosis in Adults With Compensatory Forefoot Varus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: effected by the epidemic of COVID-19
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM108087F
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Forefoot Varus; Flat Feet
Keywords: Forefoot varus; Forefoot medial wedge; Flat foot; Orthoses
MeSH Terms: conditions — Metatarsus Varus; Flatfoot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arch support orthoses with forefoot medial wedge (Experimental): The intervention of this group include orthoses with arch support and added forefoot medial wedge.
  Interventions: Other: Arch support orthoses with forefoot medial wedge
- Arch support orthoses (Experimental): The intervention of this group include orthoses with arch support.
  Interventions: Other: Arch support orthoses
- Flat insole (Sham Comparator): This group will wear a flat insole. It is made from ethylene-vinyl acetate copolymer with 4mm thickness. It only provide shock absorbtion.
  Interventions: Other: Flat insole

INTERVENTIONS:
Other: Arch support orthoses with forefoot medial wedge — The degree of forefoot wedge will be 3 degree. If needed, it could be adjusted. The subjects need to wear the orthoses for at least 30 hour per week during the experiment.
  Other Names: Forefoot medial wedge
  Arms: Arch support orthoses with forefoot medial wedge
Other: Arch support orthoses — The arch support of the orthoses could be adjusted depends on the evaluation of subject. The subjects need to wear the orthoses for at least 30 hour per week during the experiment.
  Arms: Arch support orthoses
Other: Flat insole — The flat insole used as a placebo intervention. The shape of this insole is flat, and made by soft EVA. It only provide shock absorbtion without any support. The subjects need to wear the orthoses for at least 30 hour per week during the experiment.
  Arms: Flat insole

SUMMARY:
Forefoot varus is a type of foot deformities. It is asociate with subtalar joint hyperpronation, and cause too much stress over tissues around foot and lower leg during weight bearing activities.

One of the common interventions for forefoot varus is to use foot orthosis with medial forefoot wedge to accommodate the forefoot deformity. Forefoot varus has been considered as an osseus deformity and caused by insufficient talar torsion during development. However, recent studies have reported forefoot varus may not be an osseus deformity. They might be a result of soft tissue adaption. For example, subtalar joint hyperpronation and ankle equinus could lead to forefoot supination/compensatory forefoot varus, which could be mistaken for osseus forefoot varus after a long period of time. If compensatory forefoot varus is caused by soft tissue adaptions, these adaptions may have a chance to reverse.

Nowadays, orthoses which applying medial forefoot wedge to accommodate the deformity for forefoot varus deformity, and the other type orthoses which applying rearfoot medial wedge and arch support are both used in subject with forefoot varus deformity.

However, some colleges claims that using medial forefoot wedge to accommodate the deformity of forefoot varus, the deformity may be fixed after a long-term period. However, there were no studies compare the effect of arch support orthosis that with and without medial forefoot wedge.

DETAILED DESCRIPTION:
Forefoot varus is a type of foot deformities. It is asociate with subtalar joint hyperpronation, and cause too much stress over tissues around foot and lower leg during weight bearing activities.

One of the common interventions for forefoot varus is to use foot orthosis with medial forefoot wedge to accommodate the forefoot deformity. Forefoot varus has been considered as an osseus deformity and caused by insufficient talar torsion during development. However, recent studies have reported forefoot varus may not be an osseus deformity. They might be a result of soft tissue adaption. For example, subtalar joint hyperpronation and ankle equinus could lead to forefoot supination/compensatory forefoot varus, which could be mistaken for osseus forefoot varus after a long period of time. If compensatory forefoot varus is caused by soft tissue adaptions, these adaptions may have a chance to reverse.

Nowadays, orthoses which applying medial forefoot wedge to accommodate the deformity for forefoot varus deformity, and the other type orthoses which applying rearfoot medial wedge and arch support are both used in subject with forefoot varus deformity.

However, some colleges claims that using medial forefoot wedge to accommodate the deformity of forefoot varus, the deformity may be fixed after a long-term period. However, there were no studies compare the effect of arch support orthosis that with and without medial forefoot wedge.

In consideration of few studies have been done for investigating the effects of different orthoses in subjects with flat foot combined forefoot varus. Thus, the purpose of this study is to investigate the effect of different foot orthoses designs on improving pain, muscle activity and displacement of center of pressure. We hypothesized that both orthoses will have the better effect on improving pain than placebo orthoses ,and muscle activity and displacement of center of pressure of arch support orthoses group will have change which close to normal foot.

ELIGIBILITY:
Inclusion Criteria:

* Flexible flatfoot
* Angle of forefoot varus > 6 degree
* Feel leg or foot pain when walking or exercising, and pain visual analogue scale > 3 points
* The duration of wearing shoes > 30 he per week

Exclusion Criteria:

* Rigid flatfoot
* Leg length discrepancy > 1cm
* Angle of Hallux valgus > 20 degree
* With any nerve problem or disease
* Used to have trauma over lower limbs
* Had any severe joint deformity or osteoarthritis over lower limbs
* Had any acute injury (in two weeks and inflammation)
* Had wearing insole for 6 months
* Can't follow order

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Foot function index | Baseline
  This questionnaire includes 23 questions. These questions are about how difficult or pain over foot when subjects doing some functional activities.
Foot function index | 6-week intervention
  This questionnaire includes 23 questions. These questions are about how difficult or pain over foot when subjects doing some functional activities.
Pain visual analogue scale (VAS) | Baseline
  The scale is from 0 to 10 points. Zero means no pain, and ten points means extremely painful over subject's foot or leg.
Pain visual analogue scale (VAS) | 6-week intervention
  The scale is from 0 to 10 points. Zero means no pain, and ten points means extremely painful over subject's foot or leg.
Change From Baseline in Global Rating of Change Scale (GROC) | change from baseline at 6 weeks later
  To measure improvements in a patient's condition. The minimum value is -7 and it means a very great deal worse. The maximum values is +7 and it means a very great deal better.

SECONDARY OUTCOMES:
Displacement of center of force of gait cycle (medial-lateral and anterior-posterior) | Baseline and after 6-week intervention
  To determine the displacement of Cof during ambulation. We use F-Scan In-Shoe system to determine dynamic pressure, force and timing information. And to calculate the displacement of center of force of each gait cycle.
Muscle activity of tibialis anterior muscle, peroneal longus and abductor hallucis brevis | Baseline and after 6-week intervention
  Muscle activity during ambulation and single leg standing. We use electromyography to record muscle activity of tibialis anterior muscle, peroneal longus and abductor hallucis brevis.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, PhD, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming University
Locations (1):
- National Yang Ming University, Taipei, Taiwan